CLINICAL TRIAL: NCT00354770
Title: A Double-Blind, Placebo-Controlled Study of N-Acetyl Cysteine in Trichotillomania
Brief Title: N-Acetyl Cysteine in Trichotillomania
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0604M85110
Record Dates: First submitted 2006-07-18; First posted 2006-07-20 (Estimated); Results first posted 2014-01-15 (Estimated); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Trichotillomania
Keywords: Trichotillomania; Hair-pulling
MeSH Terms: conditions — Trichotillomania | interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- N-Acetyl Cysteine (Active Comparator): N-Acetyl Cysteine
  Interventions: Drug: N-Acetyl Cysteine
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — daily
  Arms: 2
Drug: N-Acetyl Cysteine — 600mg capsules in varying doses for 12 weeks.
  Other Names: NAC
  Arms: N-Acetyl Cysteine

SUMMARY:
This is a 12-week, double-blind study of N-Acetyl Cysteine in the treatment of trichotillomania

DETAILED DESCRIPTION:
The goal of the proposed study is to evaluate the efficacy and safety of N-Acetyl Cysteine (NAC) in trichotillomania. Forty subjects with DSM-IV trichotillomania will receive 12 weeks of double-blind NAC or placebo. The hypothesis to be tested is that NAC will be effective and well tolerated in patients with trichotillomania compared to placebo. The proposed study will provide needed data on the treatment of a disabling disorder that currently lacks a clearly effective treatment.

ELIGIBILITY:
Inclusion Criteria:

* men and women age 18-65;
* current DSM-IV trichotillomania

Exclusion Criteria:

* unstable medical illness;
* history of seizures;
* myocardial infarction within 6 months;
* current pregnancy or lactation, or inadequate contraception in women of childbearing potential;
* any thoughts of suicide;
* lifetime history of DSM-IV bipolar disorder type I, dementia, or schizophrenia or any other DSM-IV psychotic disorder;
* previous treatment with N-Acetyl Cysteine;
* treatment with investigational medication or depot neuroleptics within 3 months, with fluoxetine within 6 weeks, or with other psychotropics within 2 weeks prior to study baseline;
* 9) diagnosis of asthma

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2006-07; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jon E Grant, MD, JD, Principal Investigator — University of Minnesota
Locations (1):
- University of Chicago Medical Center, Chicago, Illinois, United States

REFERENCES:
- [Derived] Hoffman J, Williams T, Rothbart R, Ipser JC, Fineberg N, Chamberlain SR, Stein DJ. Pharmacotherapy for trichotillomania. Cochrane Database Syst Rev. 2021 Sep 28;9(9):CD007662. doi: 10.1002/14651858.CD007662.pub3. PMID 34582562
- [Derived] Odlaug BL, Chamberlain SR, Harvanko AM, Grant JE. Age at onset in trichotillomania:clinical variables and neurocognitive performance. Prim Care Companion CNS Disord. 2012;14(4):PCC.12m01343. doi: 10.4088/PCC.12m01343. Epub 2012 Jul 19. PMID 23251869
- [Derived] Grant JE, Odlaug BL, Kim SW. N-acetylcysteine, a glutamate modulator, in the treatment of trichotillomania: a double-blind, placebo-controlled study. Arch Gen Psychiatry. 2009 Jul;66(7):756-63. doi: 10.1001/archgenpsychiatry.2009.60. PMID 19581567

RESULTS

PARTICIPANT FLOW:
Groups:
- N-Acetyl Cysteine: N-Acetyl Cysteine (NAC) - 1200mg-2400mg by mouth per day
- Placebo: Placebo pills
Period: Overall Study
Arm/Group | N-Acetyl Cysteine | Placebo
Started | 25 | 25
Completed | 22 | 22
Not Completed | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | N-Acetyl Cysteine | Placebo | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 25 | 25 | 50
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.8 (13.6) | 32.7 (10.5) | 34.5 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 21 | 45
  Male | 1 | 4 | 5
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: Massachusetts General Hospital Hairpulling Scale
Description: There is no minimum or maximum score to quantify 'good' or 'poor' improvement based on this scale. The total score can range from 0-28 with zero being no problems to 28 being the most severe score one can receive.A total of 6 assessments were made, however only the final score (the score at the final visit after 12 weeks) was reported here to show the final outcome measure that was used in the final report of possible improvement and what was reported for final publication of data.
Time Frame: Baseline and final visit after 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | N-Acetyl Cysteine | Placebo
Number analyzed (Participants) | 25 | 25
units on a scale
  MGH-HPS Baseline | 17.6 (4.64) | 16.7 (5.28)
  MGH-HPS Final Visit After 12 Weeks | 10.4 (5.55) | 16.0 (4.90)

ADVERSE EVENTS:
Arm/Group | N-Acetyl Cysteine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 3/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | N-Acetyl Cysteine (N=25) | Placebo (N=25)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No